CLINICAL TRIAL: NCT02731755
Title: Acute Cardiovascular Effects of Phenolic Rich Oats in Men With Above Average Blood Pressure
Brief Title: Phenolic-rich Oats and Artery Improvement
Acronym: PROGRAIN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Rothamsted Research (Unknown); PepsiCo Global R&D (Industry); University of Roehampton (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PROGRAIN2
Record Dates: First submitted 2016-02-09; First posted 2016-04-08 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy
Keywords: Oats; Phenolic acid; FMD; LDI; Avenanthramide
MeSH Terms: interventions — Ornithine-Oxo-Acid Transaminase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oat intervention (Active Comparator): 67.7g oatflake and 22.5g oatbran concentrate - single intake (mixed with water)
  Interventions: Other: Oat
- Control (Placebo Comparator): 39.4g cream of rice, 6.1g sunflower oil, 29.5g skimmed milk, 5.6g pectin powder, 6.5g cellulose and mixed with water
  Interventions: Other: Control

INTERVENTIONS:
Other: Oat — The study oat intervention products will consist of 67.7g oatflake and 22.5g oatbran concentrate.
  Arms: Oat intervention
Other: Control — 60g cream of rice
  Arms: Control

SUMMARY:
In this proposed human trial, the investigators aim to establish whether consumption of one portion of phenolic acid-rich oats leads to acute improvements (i.e. 1-24h post-intake) in markers of cardiovascular disease risk relative to an energy matched control intervention in healthy men with high-normal to mildly elevated blood pressure.

DETAILED DESCRIPTION:
A diet rich in whole grain is inversely associated with cardiovascular disease risk. Whole grains contain a wide range dietary components including potentially vasoactive phenolic acids.

ELIGIBILITY:
Inclusion Criteria:

* Above average blood pressure (i.e. systolic 120-159 mmHg and diastolic 75-99 mmHg)

Exclusion Criteria:

* Abnormal biochemical, haematological results as assessed at health screening
* Hypertension (i.e. systolic/diastolic blood pressure ≥160/100 mm Hg) BMI >35
* Current smoker or ex-smoker ceasing <3 months ago
* Past or existing medical history of vascular disease, diabetes, hepatic, renal, gastrointestinal, haematological, neurological, thyroidal disease or cancer
* Prescribed or taking lipid lowering, antihypertensive, vasoactive (e.g. Viagra), anti-inflammatory, antibiotic or antidepressant medication
* Allergies to whole grains
* Parallel participation in another research project
* Having flu vaccination or antibiotics within 3 months of trial start
* On a weight reduction regime or taking food supplements within 3 months of trial start
* Performing high level of physical activity (i.e. >3 x 20 min aerobic exercise/week)
* Consumption of ≥21 units of alcohol/week
* Small veins not allowing cannulation

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with above average blood pressure
Enrollment: 18 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Spencer, Professor, Principal Investigator — University of Reading
Locations (2):
- United Kingdom (2):
  - Hugh Sinclair Unit of Human Nutrition, Reading, Berkshire
  - Hugh Sinclair Unit of Human Nutrition, Reading

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oat Then Control: The first intervention is oat, the second intervention is control
- Control Then Oat: The first intervention is control, the second intervention is oat
Period: First Intervention
Arm/Group | Oat Then Control | Control Then Oat
Started | 8 | 10
Completed | 8 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Intervention
Arm/Group | Oat Then Control | Control Then Oat
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participant: Crossover study - All participant
Arm/Group | All Participant
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 133.9 (2.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 81.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilatation
Description: Technique to assess the flexibility of the endothelium in larger peripheral blood vessels
Time Frame: 1 hour, 6 hours and 24 hours
Population: Excluded data from 2 volunteers as their results were out of the normal range
Measure: Mean (Standard Error); unit: metre
Groups:
- Oat Intervention: The first intervention is oat, the second intervention is control
- Control: The first intervention is control, the second intervention is oat
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 14 | 14
metre
  1h | 4.4 (0.7) | 3.9 (0.9)
  6h | 3.4 (0.6) | 4.4 (0.8)
  24h | 4.4 (0.4) | 3.6 (0.7)
Statistical Analysis 1: Comparison: Oat Intervention vs Control; Between time points and treatments, calculated p value; Test type: Superiority; p = 0.5, Mixed Models Analysis

2. Secondary Outcome: Laser Doppler Iontophoresis
Description: Acute postprandial timecourse from Baseline to 2 hours, 24hours, AUC - area under the blood flow and time curve Ach-iAUC-endothelium dependent incremental area under the curve SNP-iAUC-endothelium independent incremental area under the curve Ach-AUC- endothelium dependent area under the curve
Time Frame: Baseline(BL), 2hours and 24hours
Population: Excluded data from 2 volunteers as their results were out of the normal range
Measure: Mean (Standard Error); unit: PU per hour
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 14 | 14
PU per hour
  Ach-i AUC, BL | 538.2 (90.4) | 465 (70.6)
  Ach-i AUC, 2h | 681.8 (182) | 463.7 (55.4)
  Ach-i AUC, 24h | 381.3 (61.4) | 315 (45.5)
  SNP-iAUC BL | 661.1 (52.4) | 757.1 (43.2)
  SNP-iAUC 2h | 709.4 (68.4) | 502.9 (25.6)
  SNP-iAUC,24h | 622.4 (50.6) | 513.7 (35.8)
  Ach-AUC, BL | 1593.9 (198.9) | 1534.1 (144.2)
  Ach-AUC, 2h | 1678.3 (140.6) | 1358.3 (116.9)
  Ach-AUC, 24h | 1560.9 (161.3) | 1701.6 (190.9)
Statistical Analysis 1: Comparison: Oat Intervention vs Control; Ach-iAUC; Test type: Superiority; p = 0.04, Mixed Models Analysis
Statistical Analysis 2: Comparison: Oat Intervention vs Control; SNP-IAUC; Test type: Superiority; p = 0.007, Mixed Models Analysis
Statistical Analysis 3: Comparison: Oat Intervention vs Control; Ach - AUC; Test type: Superiority; p = 0.02, Mixed Models Analysis

3. Secondary Outcome: Phenolic Acids Metabolites - Ferulic Acid
Description: Concentration of phenolic acid metabolites in plasma and urine as Assessed by liquid chromatography/mass spectrometry magnitude of increase from Baseline to 24h
Time Frame: Baseline, 1hour, 2 hours and 24hours
Population: Excluded data from 2 volunteers as their results were out of the normal range
Measure: Mean (Standard Deviation); unit: nanomolars
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 14 | 14
nanomolars
  BL | 10.6 (7.8) | 0.4 (2.4)
  1h | 33.9 (17.5) | 9 (6.4)
  2h | 153.5 (145.2) | 10.3 (9.3)
  24h | 373 (4) | 222 (24)
Statistical Analysis 1: Comparison: Oat Intervention vs Control; Test type: Superiority; p = 0.9, Mixed Models Analysis

4. Secondary Outcome: Plasma Nitric Oxide Analysis
Description: Concentration of nitric oxide in nmol
Time Frame: Acute postprandial timecourse from Baseline, 1hour to 24hours.
Population: No data collected
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: NADPH Oxidase Activity in Neutrophil Blood Cells
Description: NADPH oxidase activity will be calculated as the difference between values obtained in PMA The fluorescence intensity was measured by C6 Flow Cytometer
Time Frame: Baseline, 2 hours and 24 hours
Population: Excluded data from 2 volunteers as their results were out of the normal range
Measure: Mean (Standard Error); unit: fluorescence intensity
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 14 | 14
fluorescence intensity
  BL | 55.7 (7) | 58.6 (8)
  2h | 43.6 (5) | 47.9 (8)
  24h | 63.6 (6) | 61.6 (9)
Statistical Analysis 1: Comparison: Oat Intervention vs Control; Test type: Superiority; p = 0.7, Mixed Models Analysis

6. Secondary Outcome: Plasma Glucose
Description: Glucose concentration in mmol/L
Time Frame: Acute postprandial timecourse from Baseline, 1hour to 24hours.
Population: Data not collected
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Plasma Insulin
Description: Insulin concentration in pmol/L
Time Frame: Acute postprandial timecourse from Baseline, 1hour to 24hours.
Population: Data not collected
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Renin Activity
Description: Renin activity in ng/(mL*hour)
Time Frame: Acute postprandial timecourse from Baseline, 1hour to 24hours.
Population: Data not collected
Arm/Group | Oat Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Oat Intervention: Participants received oat intervention
- Control: Participants received control intervention
Arm/Group | Oat Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oat Intervention (N=18) | Control (N=18)
Faint (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes